CLINICAL TRIAL: NCT01763372
Title: Functional Implications of Arthroscopic Iliopsoas Release
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stephen Aoki, M.D., University of Utah
Other Study IDs: 58424
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Arthroscopic Iliopsoas Release
Keywords: Arthroscopic; Iliopsoas; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the functional effects of arthroscopic iliopsoas release. To complete this aim, we will recruit patients who have undergone arthroscopic iliopsoas release by Dr. Aoki. Each subjects contralateral nonoperative hip will serve as their own control. To delineate the effects of arthroscopic surgery alone from those resulting from iliopsoas release in addition to arthroscopic surgery, we will recruit a second control group consisting of patients who have undergone arthroscopic surgery by Dr. Aoki without iliopsoas release.

For both hips of each subject, we will:

* Quantify the muscle volume of the iliopsoas muscle with MRI.
* Quantify hip flexion strength with isokinetic dynamometry.
* Quantify patient function and satisfaction with functional outcome surveys.

This data will allow us to test the following hypotheses:

* Compared to the non-operative hip, hips undergoing arthroscopic iliopsoas release have decreased iliopsoas muscle volume and hip flexion strength.
* Compared to hips undergoing arthroscopic surgery without iliopsoas release, hips undergoing arthroscopic iliopsoas release have decreased iliopsoas muscle volume and hip flexion strength.
* Patient function and satisfaction positively correlates to muscle bulk and strength.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be greater than 18 years of age.
* We will recruit 18 subjects who have undergone arthroscopic iliopsoas release by Dr. Aoki.
* We will recruit 18 additional subjects that had hip arthroscopy with Dr. Aoki without iliopsoas release to serve as a control group.

Exclusion Criteria:

* As the nonoperative contralateral hip will serve as a control to the operative hip, we will exclude patients for this study who have undergone bilateral procedures.
* We will exclude any patients who are not comfortable with the MRI scan, stationary bike or strength testing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing arthroscopic surgery by Dr. Aoki, divided into two groups:
  Those undergoing arthroscopic psoas release, and those undergoing arthroscopic surgery without psoas release,
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Muscle Volume | 1 yr post op

SECONDARY OUTCOMES:
Hip Flexion Strength | 1 yr post op

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aoki, Principal Investigator — Orthopedic Surgery Operations